CLINICAL TRIAL: NCT00873405
Title: Banded Sleeve Gastrectomy Versus Banded Ring Gastric Bypass in Morbidly Obese Patients: a Prospective Controlled Trial.
Brief Title: Banded Sleeve Gastrectomy Versus Banded Ring Gastric Bypass in Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Gustavo Peixoto Soares Miguel, Federal University of Espirito Santo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 049/06
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: Type 2 diabetes mellitus; Metabolic control; Bariatric Surgery; Weight Loss; Sleeve gastrectomy; BMI reduction; Waist circumference reduction; Percentage of excess BMI loss; Glucose homeostasis
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRSG (Active Comparator): Silastic® ring sleeve gastrectomy (SRSG).
  Interventions: Procedure: Silastic® ring sleeve gastrectomy
- SRGB (Other): Silastic® ring gastric bypass.
  Interventions: Procedure: Silastic® ring sleeve gastrectomy; Procedure: Silastic® ring gastric bypass

INTERVENTIONS:
Procedure: Silastic® ring sleeve gastrectomy — SRSG group: ligation of the vessels of the greater curvature of the body and fundus of stomach; resection of the fundus and part of the body of stomach using a linear stapler (80 mm, Tyco®) and a 32-Fr tube to calibrate the remaining stomach; placement of a 6.2 cm Silastic® ring around the stomach, 5.0 cm below the esophagogastric junction.
  Other Names: Sleeve gastrectomy
Procedure: Silastic® ring gastric bypass — SRGB group: creation of a small, proximal gastric pouch using a linear stapler (80 mm, Tyco®) and a 32-Fr tube to calibrate the gastric pouch; creation of an intestinal loop of 150 cm and a biliopancreatic loop of 40 cm; placement of a 6.2 cm Silastic® ring around the stomach, 5.0 cm below the esophagogastric junction.
  Other Names: gastric bypass
  Arms: SRGB

SUMMARY:
Obesity is a multifactorial disease that affects millions of people worldwide. It is the main independent risk factor for developing type 2 diabetes mellitus (T2DM). Most patients with T2DM and glucose intolerance (GI) are overweight, a condition known as diabesity. In patients with the most severe form of obesity, i.e., morbid obesity, the likelihood of developing diseases associated with obesity is increased.

The investigators currently know that bariatric surgery provides sustained weight loss and well-documented remission of T2DM. Patients who undergo bariatric surgery show long-term reduced mortality from coronary artery disease, cancer and diabetes; 136 lives are saved per 10,000 surgical procedures performed. Bariatric surgery is a relatively safe procedure that is becoming increasingly well-accepted; in 2007, approximately 170,000 bariatric procedures were performed in the USA. Currently, bariatric surgery is the most effective choice of treatment of morbidly obese patients with diabetes.

The surgical procedures that are currently performed to treat morbid obesity are divided into two main groups: gastric restrictive procedures and combination procedures; the latter combine gastric restriction and malabsorption. The roux-en-Y gastric bypass (RYGB) is the combination procedure most frequently performed, whereas sleeve gastrectomy (SG) is an emerging restrictive procedure. SG can be performed as the first of a two-stage operation in patients at high risk of death, or as a definitive surgical procedure. It has shown good results with regard to weight loss and glycemic control in various studies. The potential advantages of SG include lower probability of vitamin and mineral deficiencies because this procedure has no malabsorptive component; access to the entire intestinal tract; no need for a subcutaneous access port or adjustments; absence of dumping syndrome and lower probability of intestinal obstruction. In addition, SG can be performed in patients who have inflammatory bowel disease or who have undergone bowel surgery, and it can be easily converted into RYGB. Both SG and RYGB can be performed with or without the placement of a Silastic® ring.

The metabolic control achieved with bariatric procedures has been demonstrated and reproduced in various medical centers worldwide. Metabolic control can be achieved with gastric restrictive procedures such as vertical banded gastroplasty, adjustable gastric banding and, more recently, SG. However, it has been shown that glucose homeostasis is affected by various intestinal mechanisms observed exclusively in procedures that include a malabsorptive element, such as RYGB.

A systematic review of 22,094 cases of morbidly obese patients submitted to bariatric surgery has shown that resolution of T2DM was achieved in 76.8% of the cases, improvement being achieved in 86% of cases. Among the criteria used to diagnose metabolic syndrome, fasting glucose levels are the first to return to normal in patients submitted to Silastic® ring gastric bypass (SRGB), a modification of the traditional RYGB which consists in adding a Silastic® ring to the gastric bypass operation. Normoglycemia after bariatric procedures, as well as diabesity itself, is multifactorial. Normoglycemia is observed as a result of dietary control, decreased plasma levels of ghrelin, weight loss and reduction of body fat, as well as of the release of gastrointestinal hormones that interfere with the function of pancreatic β cells (incretins).

The main purpose of this study was to compare the weight loss of morbidly obese patients submitted to either a Silastic® ring sleeve gastrectomy (SRSG) or an SRGB, as well as to compare the effects of both procedures on glucose homeostasis in morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged 20-60 years
* BMI 40-45 (inclusive)
* agreed on giving written informed consent

Exclusion Criteria:

* secondary obesity
* alcohol or drug use
* severe psychiatric disorder
* binge-eating of sweets
* previous stomach or bowel surgery

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Weight loss, BMI reduction and waist circumference reduction | 12 months

SECONDARY OUTCOMES:
Glucose homeostasis, metabolic control. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo PS Miguel, Surgery Assistant Professor, Principal Investigator — Federal University of Espírito Santo
Locations (1):
- Cassiano Antonio Moraes University Hospital, Federal University of Espírito Santo, Vitória, Espírito Santo, Brazil

REFERENCES:
- [Background] Lee CM, Cirangle PT, Jossart GH. Vertical gastrectomy for morbid obesity in 216 patients: report of two-year results. Surg Endosc. 2007 Oct;21(10):1810-6. doi: 10.1007/s00464-007-9276-y. Epub 2007 Mar 14. PMID 17356932
- [Background] Cottam D, Qureshi FG, Mattar SG, Sharma S, Holover S, Bonanomi G, Ramanathan R, Schauer P. Laparoscopic sleeve gastrectomy as an initial weight-loss procedure for high-risk patients with morbid obesity. Surg Endosc. 2006 Jun;20(6):859-63. doi: 10.1007/s00464-005-0134-5. Epub 2006 Apr 22. PMID 16738970
- [Background] Silecchia G, Boru C, Pecchia A, Rizzello M, Casella G, Leonetti F, Basso N. Effectiveness of laparoscopic sleeve gastrectomy (first stage of biliopancreatic diversion with duodenal switch) on co-morbidities in super-obese high-risk patients. Obes Surg. 2006 Sep;16(9):1138-44. doi: 10.1381/096089206778392275. PMID 16989696
- [Background] Baltasar A, Serra C, Perez N, Bou R, Bengochea M, Ferri L. Laparoscopic sleeve gastrectomy: a multi-purpose bariatric operation. Obes Surg. 2005 Sep;15(8):1124-8. doi: 10.1381/0960892055002248. PMID 16197783
- [Background] Moon Han S, Kim WW, Oh JH. Results of laparoscopic sleeve gastrectomy (LSG) at 1 year in morbidly obese Korean patients. Obes Surg. 2005 Nov-Dec;15(10):1469-75. doi: 10.1381/096089205774859227. PMID 16354529
- [Background] Vidal J, Ibarzabal A, Romero F, Delgado S, Momblan D, Flores L, Lacy A. Type 2 diabetes mellitus and the metabolic syndrome following sleeve gastrectomy in severely obese subjects. Obes Surg. 2008 Sep;18(9):1077-82. doi: 10.1007/s11695-008-9547-2. Epub 2008 Jun 3. PMID 18521701
- [Background] Fobi M. Why the Operation I Prefer is Silastic Ring Vertical Gastric Bypass. Obes Surg. 1991 Dec;1(4):423-426. doi: 10.1381/096089291765560854. PMID 10775946
- [Background] Buchwald H, Buchwald JN. Evolution of operative procedures for the management of morbid obesity 1950-2000. Obes Surg. 2002 Oct;12(5):705-17. doi: 10.1381/096089202321019747. PMID 12448398
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Cummings DE, Overduin J, Foster-Schubert KE. Gastric bypass for obesity: mechanisms of weight loss and diabetes resolution. J Clin Endocrinol Metab. 2004 Jun;89(6):2608-15. doi: 10.1210/jc.2004-0433. No abstract available. PMID 15181031
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Langer FB, Reza Hoda MA, Bohdjalian A, Felberbauer FX, Zacherl J, Wenzl E, Schindler K, Luger A, Ludvik B, Prager G. Sleeve gastrectomy and gastric banding: effects on plasma ghrelin levels. Obes Surg. 2005 Aug;15(7):1024-9. doi: 10.1381/0960892054621125. PMID 16105401
- [Background] Nakazato M, Murakami N, Date Y, Kojima M, Matsuo H, Kangawa K, Matsukura S. A role for ghrelin in the central regulation of feeding. Nature. 2001 Jan 11;409(6817):194-8. doi: 10.1038/35051587. PMID 11196643
- [Background] Pories WJ, Albrecht RJ. Etiology of type II diabetes mellitus: role of the foregut. World J Surg. 2001 Apr;25(4):527-31. doi: 10.1007/s002680020348. Epub 2001 Apr 18. PMID 11344408
- [Background] Cai J, Zheng C, Xu L, Chen D, Li X, Wu J, Li J, Yin K, Ke Z. Therapeutic effects of sleeve gastrectomy plus gastric remnant banding on weight reduction and gastric dilatation: an animal study. Obes Surg. 2008 Nov;18(11):1411-7. doi: 10.1007/s11695-008-9490-2. Epub 2008 Apr 26. PMID 18438617
- [Background] Braghetto I, Korn O, Valladares H, Gutierrez L, Csendes A, Debandi A, Castillo J, Rodriguez A, Burgos AM, Brunet L. Laparoscopic sleeve gastrectomy: surgical technique, indications and clinical results. Obes Surg. 2007 Nov;17(11):1442-50. doi: 10.1007/s11695-008-9421-2. PMID 18219770
- [Background] Deitel M, Gawdat K, Melissas J. Reporting weight loss 2007. Obes Surg. 2007 May;17(5):565-8. doi: 10.1007/s11695-007-9116-0. No abstract available. PMID 17658011